CLINICAL TRIAL: NCT05481528
Title: A Randomized, Double-blind, Placebo- and Moxifloxacin-controlled Study to Investigate the Safety and Pharmacokinetics of Single Ascending Supratherapeutic Doses of Elinzanetant in Healthy Participants
Brief Title: A Study to Learn How Safe the Study Treatment Elinzanetant is and How it Moves Into, Through and Out of the Body When Given as Single Increasing Doses That Are Higher Than Normally Used Compared to Placebo and Moxifloxacin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 21670; 2022-000056-11 (EudraCT Number)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men; Hot Flashes; Healthy Volunteers
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Hot Flashes | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1 - Dose group 1 (Experimental): Single oral dose of elinzanetant or placebo.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo
- Part 1 - Dose group 2 (Experimental): Single oral dose of elinzanetant or placebo
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo
- Part 1 - Dose group 3 (Experimental): Single oral dose of elinzanetant or placebo
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo
- Part 1 - Dose group 4 (Experimental): Single oral dose of elinzanetant or placebo
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo
- Part 2: Moxifloxacin - Placebo (Experimental): Participants of Dose Groups 1 and 4 will receive a single dose of moxifloxacin in Period 1 and a single dose of placebo in Period 2.
  Interventions: Drug: Moxifloxacin; Drug: Placebo
- Part 2: Placebo - Moxifloxacin (Experimental): Participants of Dose Groups 1 and 4 will receive a single dose of placebo in Period 1 and a single dose of moxifloxacin in Period 2.
  Interventions: Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: Moxifloxacin — Single oral dose of 400 mg moxifloxacin
  Arms: Part 2: Moxifloxacin - Placebo; Part 2: Placebo - Moxifloxacin
Drug: Elinzanetant (BAY3427080) — Single oral dose of elinzanetant
  Arms: Part 1 - Dose group 1; Part 1 - Dose group 2; Part 1 - Dose group 3; Part 1 - Dose group 4
Drug: Placebo — Single oral dose of placebo

SUMMARY:
Researchers are looking for a better way to treat vasomotor symptoms, a condition of having hot flashes. The condition is caused by hormonal changes and occurs primarily in women, but can also affect men.

The study treatment, elinzanetant, is under development to treat symptoms caused by hormonal changes. It works by blocking a substance called neurokinin from sending signals to other parts of the body, which is thought to play a role in starting hot flashes.

Participants of this study will be healthy and will have no benefit from administration of elinzanetant. This study, however, will provide information on how to use it in people with vasomotor symptoms.

In previous studies, elinzanetant doses tested and resulting blood levels were close to the levels intended for treatment. However, in future use, it cannot always be ruled out that higher elinzanetant concentrations may occur in the blood if patients are taking certain other drugs at the same time, or take more than the recommended dose of the drug.

The main purpose of this study is to learn how safe elinzanetant is when higher doses than normally used are given compared to placebo in healthy participants. A placebo is a treatment that looks like a medicine but does not have any medicine in it.

To answer this, researchers will compare the number of participants who have medical problems after taking elinzanetant to those treated with placebo. Doctors keep track of all medical problems that happen in studies, even if they do not think they might be related to the study treatments.

The study consists of two parts. In part 1, the participants will either take a single dose of elinzanetant or placebo by mouth dependent on the treatment group. Four different increasing doses of elinzanetant will be tested.

Participants in dose group 1 and 4 will participate in part 2. About 8 days after treatment in part 1, the participants will receive a single dose of moxifloxacin and a single dose of placebo as tablet by mouth 5 days apart. Whether the participant starts with moxifloxacin or placebo is decided by chance. Moxifloxacin is used to make sure that certain changes in heart rhythm can be detected in the study.

Each participant will be in the study for about 6 weeks including 1 treatment day (part 1) or for about 8 weeks including 3 treatment days (part 1 & 2). Participants of part 1 will stay in-house for 7 days. Participants of part 2 will stay in-house for another 9 days. The in-house phase starts two days before intake of the study treatment. In addition, one visit before and one visit after the in-house phase to the study site is planned.

During the study, the study team will:

* Do physical examinations
* Check vital signs
* Take blood and urine samples
* Examine the participants' heart health using electrocardiogram (ECG)
* Ask the participants questions about their mood and about sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, blood pressure, pulse rate, respiratory rate, body temperature and electrocardiogram (ECG).
* Body weight of at least 50 kg.
* Body mass index (BMI) within the range 18.0 to 30.0 kg/m^2 (inclusive).
* Male subjects of reproductive potential must agree to use a condom (with or without spermicide) when sexually active with a female partner and refrain from donating sperm. This applies for the time period between the signing of the informed consent form (ICF) until 5 days after the last administration of study intervention. Female partners of childbearing potential of male subjects do not need to follow special precautions.
* Women of childbearing potential will have to use a highly effective non-hormonal contraception when having sexual intercourse with a male partner from signing of the ICF until 5 days after the last administration of study intervention.

Exclusion Criteria:

* Any clinically relevant abnormal findings in medical history and physical examination. Including: History or evidence of any clinically relevant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other clinically relevant disease, as judged by the investigator; Diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention will not be normal.
* Known or suspected hypersensitivity or allergy to the study interventions or other fluoroquinolone products.
* Relevant diseases within the last 4 weeks prior to the first administration of study intervention, including febrile illness.
* Contraindications for the use of moxifloxacin, including: Medical history of seizures or psychiatric disorders, myasthenia gravis, severe cutaneous adverse reactions (SCARs) including toxic epidermal necrolysis (TEN; also known as Lyell's syndrome), Stevens Johnson syndrome (SJS) and Acute Generalized Exanthematous Pustulosis (AGEP), glucose-6-phosphate dehydrogenase deficiency.
* Pregnant or breastfeeding women.
* Tendency for vasovagal reactions or history of syncope.
* Use of mild, moderate, or strong CYP3A4 and P-gp inhibitors from 2 weeks, and use of CYP3A4 and P-gp inducers from 4 weeks prior to the first administration of study intervention.
* Use of drugs which may affect absorption and systemic administration of any broad-spectrum antibiotic within 1 week prior to first administration of study intervention.
* Use of drugs which may affect absorption by increasing the gastrointestinal pH e.g. proton pump inhibitors from 2 weeks prior to first administration of study intervention.
* Use of any herbal products or St. John's wort within 4 weeks prior to the first administration of study intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and severity of TEAEs related to elinzanetant | After first application of study intervention until 20 days after last application of study intervention

SECONDARY OUTCOMES:
AUC (if AUC cannot be determined reliably in all subjects, AUC(0-tlast) will be used instead) of elinzanetant | 0 - 96 hours post-dose
  AUC stands for area under the concentration versus time curve from zero to infinity
Cmax of elinzanetant | 0 - 96 hours post-dose
  Cmax stands for maximum observed concentration

CONTACTS AND LOCATIONS:
Locations (1):
- NUVISAN GmbH Neu-Ulm, Neu-Ulm, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.